CLINICAL TRIAL: NCT00175422
Title: The Period of PURPLE Crying: An Educational Intervention to Change the Knowledge, Attitudes and Behaviour of New Parents About Early Infant Crying
Brief Title: Parents Helping Infants Study: Educational Intervention to Change the Knowledge, Attitudes and Behaviour of New Parents About Early Infant Crying
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Ronald Barr, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B04-0785
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Shaken Baby Syndrome
Keywords: Prevention; Randomized controlled trial; Community education; Shaken Baby Syndrome; Crying; Colic
MeSH Terms: conditions — Shaken Baby Syndrome; Health Education; Crying; Colic

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Behavioral: The Period of PURPLE Crying Program — There are two treatment arms in the study. The first half of all subjects (n=500) will receive the PURPLE intervention materials (a video and a pamphlet) about infant crying. The second arm will receive comparable materials on infant safety and SIDS.

SUMMARY:
This research project seeks to implement an early intervention program that can be effective in the prevention of shaken baby syndrome (SBS) and infant abuse. The investigators' hypothesis is that the Period of PURPLE Crying intervention program can be effective in reducing the shaking and abuse of infants through changes in knowledge, attitudes and behaviours about early infant crying, especially inconsolable crying.

DETAILED DESCRIPTION:
The Period of PURPLE Crying phrase refers to the educational information and the action steps that caregivers need to know about the properties of early crying in normally developing infants that are uniformly frustrating to caregivers. The study will be implemented and evaluated in 1000 new mothers, by public health nurses during newborn home care visits in the Vancouver Coastal and Fraser Health Authorities. There are two treatment arms in the study. The first half of all subjects (n=500) will receive the PURPLE intervention materials (a video and a pamphlet) about infant crying. The second arm will receive comparable materials on infant safety and SIDS.

Specific goals of the research program are:

1. To change the understanding (i.e knowledge and attitudes) and reduce the frustration of parents of new infants about the normality of the frustrating properties of crying;
2. To change the behaviour of parents to increase care giving contact in response to crying but to 'walk away' if frustrated or angry;
3. To provide parents with the ability to educate other caregivers (relatives, baby sitters) to reduce frustration induced by inconsolable crying and obtain help if needed;
4. To provide parents with the knowledge to protect their infants from occasional caregivers who could harm their infants because of the frustrating nature of early crying;
5. To provide effective knowledge, skills and teaching materials to regional health care providers in direct contact with parents concerning crying, shaking and abuse.

ELIGIBILITY:
Inclusion Criteria:

* New mothers of healthy infants born at > 34 weeks gestation with access to a video or DVD player.

Exclusion Criteria:

* Mothers of: infants born at < 34 weeks gestation; multiple infants (twins, triplets, etc.); or infants who have serious medical conditions.
* Mothers who don't speak and read English.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1833 (Actual)
Dates: Start 2005-05; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To demonstrate the effectiveness of the Period of PURPLE Crying program to change knowledge, attitudes and behavior about early infant crying and shaken baby syndrome in new parents at two months of life | Two months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Barr, MD, Principal Investigator — University of British Columbia
Locations (1):
- Centre for Community Child Health Research, BC Childrens and Women's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Barr RG, Barr M, Fujiwara T, Conway J, Catherine N, Brant R. Do educational materials change knowledge and behaviour about crying and shaken baby syndrome? A randomized controlled trial. CMAJ. 2009 Mar 31;180(7):727-33. doi: 10.1503/cmaj.081419. Epub 2009 Mar 2. PMID 19255065